CLINICAL TRIAL: NCT06206018
Title: Patient-Reported Outcome Measures in Lower Extremity Rehabilitation Program PROM_R: Impact on Health Care
Acronym: PROM_R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, José Manuel Afonso Moreira, MsC, University of Évora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE-ENSP 3/2022
Record Dates: First submitted 2024-01-03; First posted 2024-01-16 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-04

CONDITIONS: Lower Extremity Problem; Rehabilitation; Knee Injuries
Keywords: Quality of Life; Patient-Reported Outcome Measures
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROM_R Knee (Experimental): Completed a rehabilitation program based on the updated Journal of Orthopaedic and Sports Physical Therapy (JOSPT) guidelines for knee injuries. These guidelines essentially refer to lower limb massage, mobilization, neuromuscular strengthening and rehabilitation, exercise literacy, neuromuscular electrical stimulation and cryotherapy.
  The intervention group will complete the four-week rehabilitation program, with five sessions per week, performed and supervised by the physiotherapist.
  Interventions: Procedure: PROM_R knee rehabilitation program
- Crontrol Group (No Intervention): The control group will follow a standard six-week rehabilitation program.

INTERVENTIONS:
Procedure: PROM_R knee rehabilitation program — The rehabilitation program consists of 5 weekly sessions for 4 weeks, supervised by a specialized physiotherapist at every session.
  All patients follow the same order of treatment and exercises, starting with massage and mobilization, followed by the corresponding exercise program, and ending with Neuromuscular Electrical Stimulation (NMES) and cryotherapy.
  Arms: PROM_R Knee

SUMMARY:
Different musculoskeletal conditions affect people all over the world and were considered by the WHO to be the leading cause of disability in 4 out of 6 regions in 2017, with an increase in the associated burden and impact on society expected in the coming years.

The knee is a complex joint, vulnerable to various types of injury. The most common are ligament, meniscus and cartilage injuries of different etiologies.

After surgery, as a result of the reflex inhibition of motor neurons and immobilization, there is rapid atrophy and weakness in the different associated muscles, affecting proprioception, muscle strength and extension, clearly compromising health-related quality of life.

Through partnership and collaboration between health institutions and academia, the rehabilitation program will take place on an outpatient basis in a supervised manner, allowing its effectiveness to be assessed using Patient-Reported Outcome Measures. These instruments are a rapidly developing topic and it is essential to understand whether the Patient-Reported Outcome Measures used are sufficient to measure the results perceived by patients with lower limb pathology who take part in rehabilitation programs.

The different Patient-Reported Outcome Measures will be applied before and after the program.

DETAILED DESCRIPTION:
The study design is a clinical trial with longitudinal assessment, with a convenience sample. Participants who meet the inclusion criteria are invited to take part and sign an informed consent form. All participants' data is encrypted and stored with password protection, and will be deleted once the results of the study have been published.

The experimental group followed the program for 4 weeks with a treatment frequency of 5 sessions per week, performed and supervised by the same specialist physiotherapist at every session.

For the statistical analysis of the data in this study, we used the Statistical Package for Social Sciences (SPSS®) 29 software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee and ankle pathology, undergoing surgery;
* That they are going to start a rehabilitation program in two Rehabilitation Clinics in coastal and inland regions of Portugal;
* Aged between 18 and 80;
* Have signed an informed consent form.

Exclusion Criteria:

* Unconsolidated fractures;
* Previous surgeries in the ipsilateral knee;
* Partial or total amputation in upper or lower limbs;
* Permanent or temporary dysfunctions of the central or peripheral nerve system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Before the intervention, after 4-6 weeks and 6 months.
  The EuroQol scale (EQ5D) makes it possible to assess quality of life in a given pathology in the general population, presented in different domains. The visual analogue scale of this questionnaire has a score of 0-100. Higher scores mean better quality of life and lower scores indicate lower quality of life.
Hospital Anxiety and Depression Scale | Before the intervention, after 4-6 weeks and 6 months.
  Participants' anxiety and worries are also assessed. Mood disorders, weakness, worry, stress, and depression are common psychological repercussions for patients with lower extremity problem. This questionnaire is made up of 14 questions. It is subdivided into two subscales - Anxiety and Depression. Each subscale has a maximum score of 21 points and the score for each subscale is analyzed separately. Scores from 0 to 7 indicate unlikely anxiety or depression; scores from 8 to 11 indicate possible but questionable anxiety or depression; scores from 12 to 21 indicate probable anxiety or depression.
Behavioural Regulations in Exercise Questionnaire | Before the intervention, after 4-6 weeks and 6 months.
  Assessment of the different aspects of motivational regulation for exercise. It is a questionnaire that evaluates and represents the differences in the ways in which people's behaviour can be regulated and how these differences are experienced. It consists of 19 items with five Likert-type response options, where 0 is 'not true for me' and 4 is 'often true for me'. This instrument assesses the following constructs: amotivation, external, introjected and identified regulation and intrinsic motivation. The results can vary from 24 (lowest self-determination) to 20 (highest self-determination).

CONTACTS AND LOCATIONS:
Locations (1):
- National School of Public Health, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Logerstedt DS, Scalzitti DA, Bennell KL, Hinman RS, Silvers-Granelli H, Ebert J, Hambly K, Carey JL, Snyder-Mackler L, Axe MJ, McDonough CM. Knee Pain and Mobility Impairments: Meniscal and Articular Cartilage Lesions Revision 2018. J Orthop Sports Phys Ther. 2018 Feb;48(2):A1-A50. doi: 10.2519/jospt.2018.0301. PMID 29385940
- [Result] Mundermann A, Dyrby CO, Andriacchi TP. Secondary gait changes in patients with medial compartment knee osteoarthritis: increased load at the ankle, knee, and hip during walking. Arthritis Rheum. 2005 Sep;52(9):2835-44. doi: 10.1002/art.21262. PMID 16145666
- [Result] Suchomel TJ, Nimphius S, Bellon CR, Stone MH. The Importance of Muscular Strength: Training Considerations. Sports Med. 2018 Apr;48(4):765-785. doi: 10.1007/s40279-018-0862-z. PMID 29372481
- [Result] Burns DJP, Arora J, Okunade O, Beltrame JF, Bernardez-Pereira S, Crespo-Leiro MG, Filippatos GS, Hardman S, Hoes AW, Hutchison S, Jessup M, Kinsella T, Knapton M, Lam CSP, Masoudi FA, McIntyre H, Mindham R, Morgan L, Otterspoor L, Parker V, Persson HE, Pinnock C, Reid CM, Riley J, Stevenson LW, McDonagh TA. International Consortium for Health Outcomes Measurement (ICHOM): Standardized Patient-Centered Outcomes Measurement Set for Heart Failure Patients. JACC Heart Fail. 2020 Mar;8(3):212-222. doi: 10.1016/j.jchf.2019.09.007. Epub 2019 Dec 11. PMID 31838032
- [Derived] Moreira J, Joao A, Aguiar P, Raimundo A, Mesquita M, Flaminio J, Almeida M, Boto P. Health-related quality of life after rehabilitation from knee surgery in rural and urban settings: a quasi-experimental study. BMC Musculoskelet Disord. 2024 Dec 19;25(1):1027. doi: 10.1186/s12891-024-08143-0. PMID 39702069